CLINICAL TRIAL: NCT00113750
Title: A Multicenter, Single-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Induction of Immunogenicity With Different Doses of Tree MATA in Subjects Allergic to Tree Pollen
Brief Title: Induction of Immunogenicity With Different Doses of TreeMATA in Subjects Allergic to Tree Pollen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TreeMATAMPL201
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Allergoid; Specific Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: TreeMATA MPL

SUMMARY:
Tree MATA (modified pollen allergen tyrosine adsorbate) has been developed to provide pre-seasonal specific immunotherapy for patients with hypersensitivity to tree (birch, alder, and hazel) pollen. Different doses of Tree MATA will be administered and immunological changes following this treatment will be assessed.

DETAILED DESCRIPTION:
Tree MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to tree (birch, alder, and hazel) pollen.

The tree pollen extract is modified with glutaraldehyde to produce the active ingredient, an allergoid. This modification reduces the reactivity of the extract with IgE antibody, thus reducing the risk of side effects. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivities, is not seen.

MPL (Monophosphoryl Lipid A), a purified, detoxified glycolipid derived from the cell wall of Salmonella minnesota, is included in the product formulation as an adjuvant to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to a TH1-like T cell profile.

The purpose of this study is to assess specific immunological changes (IgG, IgG1, IgG4 and IgE) in allergic subjects following 2 subcutaneous injections of different doses of study medication (Tree MATA) or placebo administered 3 weeks apart. The immunological changes will be used to assess the performance of the R7 IgG reactivity assay over a range of clinically efficacious doses.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential may enter the study if they have a negative urine pregnancy test and they have been practicing adequate contraception for 3 months prior to the study and continue to do so during the study
* History of at least 1 season of moderate to severe seasonal rhinoconjunctivitis without bronchial asthma due to an IgE mediated allergy to pollen from trees
* Positive skin prick test to birch, hazel and alder pollen allergen extract
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for birch with class >= 2
* Moderate/severe allergy symptoms in the past tree season
* Spirometry at Screening demonstrates FEV1 >= 80% predicted and FEV1/FVC >= 70%.

Exclusion Criteria:

* History or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of skin prick test results
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the screening skin prick tests
* History of bronchial asthma, COPD, or other chronic condition of the lower respiratory tract
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 1
* Clinically relevant sensitivity to any common perennial allergen: house dust mites, molds, or epithelia. Subjects may be enrolled in the study if they test positive, but have no current symptoms to perennial allergens
* Clinically relevant sensitivity to summer/autumn flowering plants and grasses: Grass pollen mix, rye, plantain, orache, nettle, mugwort, bermuda grass, and ragweed. Subjects may be enrolled in the study if they test positive, but have no current symptoms to these summer/autumn allergens.
* History of auto-immune diseases or rheumatoid diseases
* Subject not allowed to receive adrenalin
* Subject has disorder of tyrosine metabolism
* Subject with diseases interfering with the immune response and have received medication, which could influence the results of this study
* Subject has acute or chronic infection
* History of anaphylaxis
* History of angioedema
* History of hypersensitivity to the excipients of the study medication
* History of immunotherapy with tree allergen extracts
* Current therapy with ß-blockers
* Currently receiving anti-allergy medication or other medications with antihistaminic activity
* Subject has a positive screening test to drugs of abuse at Visit 1
* Subject received investigational medication in a clinical research trial within the last 3 months
* Subject cannot communicate reliably with the Investigator or who are not likely to cooperate with the requirements of the study
* Subject is pregnant or lactating
* Use of prohibited medications or inadequate washout periods prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70
Dates: Start 2005-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Post-injection antibody response to birch

SECONDARY OUTCOMES:
Adverse Events (AEs)
Clinical laboratory evaluations
Vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Karl Jürgen Fischer von Weikersthal-Drachenberg, MD, Study Chair — Allergy Therapeutics
Locations (10):
- United States (10):
  - Southern California Research, Mission Viejo, California
  - San Jose Clinical Research, Inc., San Jose, California
  - Rx Research, Woodstock, Georgia
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - The Medical Center at Teaneck, Teaneck, New Jersey
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington
  - A.S.T.H.M.A., Inc., Seattle, Washington
  - Pulmonary Consultants, Tacoma, Washington